CLINICAL TRIAL: NCT01726608
Title: A Sham, Controlled, Randomised Trial to Investigate the Effects of Radiofrequency Neurotomy Using Simplicity III® on Patients With Sacroiliac Joint Pain.
Brief Title: RFN for SIJ Disease Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Reda 7869
Record Dates: First submitted 2012-11-11; First posted 2012-11-15 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Sacro Iliac Joint Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiofrequency neurotomy (Active Comparator): Active Radiofrequency Neurotomy
  Interventions: Procedure: Comparison of active versus sham radiofrequency neurotomy with Simplicity III
- Sham (Placebo Comparator): Sham radiofrequency neurotomy
  Interventions: Procedure: Comparison of active versus sham radiofrequency neurotomy with Simplicity III

INTERVENTIONS:
Procedure: Comparison of active versus sham radiofrequency neurotomy with Simplicity III

SUMMARY:
The purpose of the study is to investigate if a technique called Simplicity III® Radiofrequency Neurotomy is effective in improving the management of sacroiliac joint pain. Currently there are a variety of treatments for managing this pain but there is still some doubt as to which treatments are the most effective. Simplicity III® is one such treatment for sacroiliac joint pain and has been used in the NHS for many years. It uses electrical current to generate heat around the tip of the needle placed close to the nerves that supply the sacro-iliac joint. This heat ablates the specific nerves supplying the joint and improves pain.

The traditional method used to treat this type of pain uses multiple injections to target the nerves supplying the joint. This method is however both time consuming and the results are variable depending upon the number of injections. Therefore a new electrode, called the Simplicity III®, was developed to allow the treatment to be undertaken using fewer injections. Although this treatment has received formal approval, undergone conformity assessment and is available in certain specialist NHS centres for clinical use, there is presently limited evidence with regards to its clinical efficacy. We wish to test the effectiveness of this new device in treating sacroiliac joint pain. The best way to prove the clinical effectiveness is to compare Simplicity III® against an identical procedure where the electrode is not switched on and neither the patient nor the doctor is aware whether it was switched on. Once pain has been assessed at 3 months, those patients not receiving active treatment and remaining in pain will be offered the active treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent
2. Age: 18 - 80 years old
3. Low back pain of more than 6 months duration with a minimum pain intensity of greater than 5 out of 10 on an 11-point numerical rating scale in the 7 days preceding study entry.
4. Subjects must achieve greater than 80% reduction in pain following each diagnostic, intra-articular block. Subjects must undergo 2 blocks in total prior to randomisation.
5. Female subjects of potential childbearing age must be using adequate contraception (i.e. using oral or intramuscular contraception or an IUCD) and must have a negative urine test.
6. No vulnerable patient groups shall be recruited into this study

Exclusion Criteria:

1. Subjects who do not fulfill inclusion criteria
2. Subjects who have previously been treated by any sacroiliac joint radiofrequency neurotomy
3. Subjects who are breastfeeding
4. Contraindications to local anaesthetics and radiofrequency neurotomy as listed in their respective summary of product characteristics
5. Subjects with documented or suspected alcohol or drug abuse, or who are suspected of having an addictive personality
6. Subjects to whom any of the following apply: Major trauma to the lumbar spine in the six months preceding study entry. Infection in the lumbar spine in the six months preceding study entry
7. Subjects' known to have a condition that, in the investigator's judgment precludes entry into the study.
8. Subjects with a significant psychiatric disorder (including depression) or subjects receiving anti-psychotic medication.
9. Subjects who have received an investigational drug or have used an investigational device in the 30 days preceding study entry.
10. Subjects unable to comply with the study assessments or unable to complete the questionnaires.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 3 months

SECONDARY OUTCOMES:
Pain Intensity | 6 months
Quality of pain | 3 and 6 months
  Short Form Mcgill Pain Questionnaire
Health related Quality of life | 3 and 6 months
  Short form health survey
Anxiety and Depression | 3 and 6 months
  Hospital and Depression Scale
Functional Disability | 3 and 6 months
  Oswestry Low Back Pain Disability Questionnaire
Health related quality of life and quality-adjusted life years | 3 and 6 months
  Euro Quol EQ-5D scale
Portion of patients randomised to sham requiring rescue therapy with RFN | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Mehta, MD FRCA, Principal Investigator — Barts & The London NHS Trust; Sibtain Anwar, MA MB FRCA, Study Director — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Mehta V, Poply K, Husband M, Anwar S, Langford R. The Effects of Radiofrequency Neurotomy Using a Strip-Lesioning Device on Patients with Sacroiliac Joint Pain: Results from a Single-Center, Randomized, Sham-Controlled Trial. Pain Physician. 2018 Nov;21(6):607-618. PMID 30508988